



## "Pronti A Salpare. Studio di fattibilità sulla valutazione dell'impatto della vela come ergoterapia in pazienti con malattie rare scheletriche"

| Codice dello studio: | <u>PaS</u> |
|---|---|
| Promotore ed indirizzo: | IRCCS - Istituto Ortopedico Rizzoli Via di Barbiano 1/10 40136 Bologna Italy |
| Versione e data del protocollo: | Vers. 1.1<br>Del 22.03.2024 |
| Centro coordinatore: | SC Malattie Rare Scheletriche – IRCCS Istituto Ortopedico Rizzoli |
| Sperimentatore coordinatore: | Dott. Luca Sangiorgi<br>Telefono : 051-6366342<br>E-mail : <u>luca.sangiorgi@ior.it</u> |
| Altre strutture coinvolte | ¬SC Medicina Fisica e Riabilitativa 1 – IRCCS Istituto Ortopedico<br>Rizzoli<br>¬SC Medicina Fisica e Riabilitativa 2 – IRCCS Istituto Ortopedico<br>Rizzoli<br>¬SC Laboratorio Analisi del Movimento – IRCCS Istituto<br>Ortopedico Rizzoli<br>¬MARINANDO ODV/MARINANDO 2.0 APS ASD<br>via Covignano 238 – 47923, Rimini |
| Metodologia: | : Studio pilota interventistico monocentrico. |
| Tipo: | Tipo: No profit |
| Supporto economico: | Supporto economico: Donazione The King Baudouin Foundation United States (KBFUS) Codice progetto numero (GAAC): 2024/731019 |
| Firma del protocollo dello<br>sperimentatore principale | Confermo di avere letto il protocollo e accetto di condurre questo studio in accordo con quanto previsto dalle linee guida ICH-GCP, al protocollo e a tutta la normativa prevista Dott. Luca Sangiorgi Firma |





## INDICE

| 1. | Razionale | pag. | 3 |
|-----|---------------------------------------------|------|----|
| 2. | Obiettivi dello studio | pag. | 4 |
| 3. | Disegno dello studio | pag. | 4 |
| 4. | Risultati attesi | pag. | 5 |
| 5. | Setting dello studio | pag. | 6 |
| 6. | Popolazione | pag. | 6 |
| 7. | Variabili da rilevare e fonte | pag. | 6 |
| 8. | Tempistica | pag. | 8 |
| 9. | Analisi statistica | pag. | 8 |
| 10. | Procedura di arruolamento | pag. | 8 |
| 11. | Raccolta dati | pag. | 8 |
| 12. | Principi etici | pag. | 8 |
| 13. | Consenso informato | pag. | 9 |
| 14. | Privacy | pag. | 9 |
| 15. | Report finale e pubblicazione dei risultati | pag. | 9 |
| 16. | Finanziamento | pag. | 9 |
| 17 | Bibliografia | paa | 10 |



#### 1. RAZIONALE

Sono definite rare quelle malattie che colpiscono un numero ristretto di persone e si configurano come condizioni debilitanti a carattere cronico [1]. Secondo le stime dell'OMS, nel Mondo, gli individui con diagnosi di malattia rara sono circa 300 milioni, in Europa tra i 27 e i 36 milioni e in Italia fra 2,1 e 3,5 milioni [2,3] con evidenti ripercussioni sia a livello individuale che comunitario impattando non solo sulla persona affetta, ma coinvolgendo anche dalle sue reti di riferimento fino al sistema sociale e assistenziale nel suo insieme.

Al fine di fronteggiare le criticità scaturite dalla rarità di tali patologie, sono stati messi in atto a livello comunitario e nazionale una serie di provvedimenti [3] con l'obiettivo di favorire la realizzazione di percorsi clinico-diagnostici-trattamentali adeguati. In particolare, a livello nazionale, prima con il "Piano Nazionale Malattie Rare 2013-2016" ma soprattutto con la promulgazione del "Testo Unico sulle Malattie Rare" (L.175/2021), è prioritario lo "sviluppo di una strategia integrata, globale e di medio periodo per l'Italia sulle malattie rare, centrata sui bisogni assistenziali della persona e della sua famiglia e definita con il coinvolgimento di tutti i portatori di interesse, tenuto conto delle esperienze già maturate" con la definizione di percorsi diagnostico-terapeutici assistenziali mirati. In ottemperanza alle direttive europee, nazionali e regionali, con Delibera n. 188 del 30 luglio 2018 è stato istituito il Centro Malattie Rare Scheletriche (Ce.Ma.RS) dell'Istituto Ortopedico Rizzoli finalizzato "all'armonizzazione e messa a sistema delle expertise sulle malattie rare scheletriche presenti, attraverso l'attivazione di una rete integrata multidisciplinare volta a proporre percorsi terapeutici specifici, dando così piena realizzazione alla normativa in materia", favorendo una diagnosi tempestiva, una presa in carico adeguata, garantendo l'accessibilità alle terapie più innovative, proponendo percorsi di sostegno per promuovere l'empowerment dei pazienti e dei loro familiari ed infine facilitando una attiva collaborazione e uno scambio continuo con le associazioni dei pazienti.

L'Adventure Therapy (AT) è una terapia esperienziale che, grazie al suo approccio innovativo basato sull'esposizione alla natura dei partecipanti, si è rivelato nel corso degli anni un trattamento efficace per migliorare l'autostima, l'autonomia e le capacità relazionali di persone rese fragili da malattie rare, croniche e disabilità [4]. L'interazione fra individuo, gruppo e natura favorisce la sperimentazione del proprio concetto di sé come parte di una riabilitazione complessiva fisica, cognitiva, emotiva o sociale. Fra le differenti attività che si possono svolgere all'aria aperta, la vela è un'attività particolarmente apprezzata tra le persone con e senza disabilità, in quanto favorisce il divertimento, l'inclusione e la partecipazione [5-7]. La letteratura conferma, infatti, la validità di processi avventurosi, emotivamente significativi, costruiti in un contesto ludico relazionale intenso, sullo stato di benessere fisico e mentale dei partecipanti, soprattutto in pazienti con malattie croniche, genetiche, metaboliche e oncologiche [8-11].

Dal punto di vista riabilitativo, l'attività velica mostra risultati positivi sul funzionamento di soggetti con disabilità attraverso la dimensione delle attività (comportamenti messi in atto per svolgere mansioni ed azioni) e della partecipazione (coinvolgimento di una persona nelle situazioni di vita) secondo la Classificazione Internazionale del Funzionamento (International Classification of Functioning, OMS 2001). In particolare, la persona con disabilità che partecipa a sport ricreativi come la vela, percepisce un aumento delle capacità fisica che può tradursi in una sensazione di migliore situazione di vita [7,12].

In tale ottica, la finalità del presente studio è di valutare la fattibilità di utilizzare l'attività velica come ergoterapia in pazienti con malattie rare scheletriche, in termini di miglioramento delle capacità fisiche, cognitive e sociali.



#### 2. OBIETTIVI DELLO STUDIO

#### ¬ Obiettivo primario:

Valutare la fattibilità di implementare un programma di ergoterapia basato sull'attività nautica per migliorare le capacità fisiche, psicologiche e sociali delle persone affette da malattie rare scheletriche.

#### Obiettivi secondari:

- Valutare le variazioni individuali nella percezione di sicurezza e abilità nel compiere un movimento.
- o Valutare le variazioni individuali nella percezione del proprio valore e delle proprie capacità.
- o Valutare le variazioni individuali nella qualità di vita.
- o Identificare un set standard di parametri funzionali ed esercizi riabilitativi.

#### 3. DISEGNO DELLO STUDIO

Studio pilota interventistico e monocentrico.

Lo studio si articolerà in 4 fasi all'interno delle quali saranno svolte attività specifiche e le relative valutazioni, come riportato in Tabella 1.

Tabella 1. Fasi dello studio Pa\$

| | FASE | ATTIVITÁ | STRUMENTI D | VALUTAZIONE |
|---|---|---|---|---|
| Fase 1 | Arruolamento | 1.1 Promozione progetto<br>1.2 Arruolamento<br>1.3 Valutazione (T <sub>0</sub> ) | CORE-OM<br>PODCI<br>EQ-5D<br>RSES | Scala di Tinetti<br>Scala Berg<br>Tampa scale |
| Fase 2 | Pre-imbarco | 2.1 Formazione all'attività nautica | | |
| Fase 3 | Imbarco | <ul> <li>3.1 Valutazione pre-attività (T<sub>1</sub>)</li> <li>3.2 Attività nautica</li> <li>3.3 Debriefing e attività di recupero</li> <li>3.4 Valutazione post-attività (T<sub>2</sub>)</li> </ul> | CORE-OM<br>PODCI<br>EQ-5D<br>RSES | IMU<br>Scala di Tinetti<br>Scala Berg<br>Tampa scale |
| Fase 4 | Post-imbarco | 4.1 Valutazione follow-up (T <sub>3</sub> ) | CORE-OM<br>PODCI<br>EQ-5D<br>RSES | Scala di Tinetti<br>Scala Berg<br>Tampa scale |

CORE-OM: Clinical Outcomes in Routine Evaluation-Outcome Measure; PODCI: Pediatric Outcomes Data Collection Instrument; EQ-5D: EuroQol 5-Dimensions; RSES: Rosenberg Self-Esteem Scale; WHODAS 2.0: World Health Organisation Disability Assessment Schedule II; IMU: Inertial Motion Units

## ¬ Fase 1:

- o Promozione del progetto sia tramite associazioni dei pazienti che via social media dell'Istituto
- o Inizio-Fine arruolamento dei partecipanti presso gli ambulatori della SC Malattie Rare Scheletriche: verifica dei criteri di inclusione/esclusione dei soggetti che hanno manifestato interesse, firma del consenso informato, e valutazione (To) tramite raccolta dati, somministrazione batteria di questionari e scale funzionali.
- ¬ Fase 2:





 Realizzazione di incontro formativo via piattaforma GoTo Meeting tra gli 8 partecipanti e i loro genitori/tutori legali, nel caso di soggetti minorenni, con i responsabili dell'associazione Marinando ODV sui principi e le buone pratiche della vela

#### ¬ Fase 3:

- o I partecipanti e i loro accompagnatori saranno alloggiati presso "Palazzo Manzoni" (RA) nel periodo 27-31 maggio 2024, sede in cui verranno effettuate sia le valutazioni T<sub>1</sub> (27 maggio) che T<sub>2</sub> (31 maggio) tramite somministrazione batteria di questionari e scale funzionali, valutazione movimenti tramite IMU. Inoltre, sarà la sede degli incontri di debriefing e delle attività motorie di recupero post-attività velica quotidiani.
- o A partire dal 27 maggio pomeriggio fino al 30 maggio pomeriggio, i partecipanti e i loro accompagnatori saranno trasferiti presso il Proto turistico di Marina di Ravenna Marinara (RA) per effettuare l'attività velica in collaborazione con Marinando ODV, per un totale di 4 h/die.

#### ¬ Fase 4:

o Verrà effettuata una visita di follow-up a tre mesi di distanza presso l'ambulatorio della SC Malattie Rare Scheletrica. In tale occasione verrà effettuata la valutazione conclusiva T<sub>3</sub>. Tale valutazione avverrà tramite somministrazione batteria di questionari e scale funzionali.

Tutte le attività previste nelle quattro fasi saranno svolte dalla SC Malattie Rare Scheletriche in collaborazione con la SC Medicina Fisica e Riabilitativa 1, SC Medicina Fisica e Riabilitativa 2 e SC Laboratorio Analisi del Movimento, coerentemente con le specifiche expertise.

#### 4. RISULTATI ATTESI

A seguito dell'attività velica, i risultati attesi sono:

- Breve termine (valutazione pre-post esperienza)

| Benefici psicologici |
|---------------------------------------------------|
| Apprendimento di nuove abilità |
| Maggiore consapevolezza di sé e del proprio corpo |
| Rafforzamento del senso di fiducia in se stessi |
| e nelle proprie capacità |
| Rafforzamento della capacità di socializzare |

## Medio termine (follow-up 3 mesi)

| Benefici fisici | Benefici psicologici |
|---|---|
| Consolidamento della forza e della resistenza muscolare | Miglioramento nella capacità di affrontare le sfide |
| Consolidamento del trofismo muscolare | Stabilizzazione consapevolezza di sé e<br>del proprio corpo |
| Consolidamento della propriocezione (percezione del corpo nello spazio) | Stabilizzazione del senso di fiducia in se<br>stessi e nelle proprie capacità |
| Consolidamento del controllo posturale | Stabilizzazione della capacità di socializzare |





Consolidamento dei muscoli stabilizzatori Consolidamento della coordinazione motoria

#### 5. SETTING DELLO STUDIO

A seconda delle attività da svolgere, le sedi saranno:

- Arruolamento, Consenso Informato, prima visita e follow-up: SC Malattie Rare Scheletriche –
   IRCCS Istituto Ortopedico (Bologna) (<a href="https://www.ior.it/en/curarsi-al-rizzoli/rare-diseases">https://www.ior.it/en/curarsi-al-rizzoli/rare-diseases</a>)
- Formazione: piattaforma GoTo Meeting
- ¬ Attività velica e accomodation:
  - Marinando ODV (Marina di Ravenna), presso il porto turistico di Marina di Ravenna, Marinara (https://www.marinara.it/it/)
  - o "Palazzo Manzoni", San Zaccaria (RA) (https://www.palazzomanzoni.it/)

#### 6. POPOLAZIONE

Trattandosi di uno studio pilota di fattibilità, e data la rarità della casistica, si prevede l'inclusione di un massimo di 8 pazienti.

I pazienti selezionati dovranno soddisfare i criteri di inclusione/esclusione sotto descritti.

## ¬ Criteri di inclusione:

- Soggetti di ambo i sessi
- o Diagnosi clinica e/o molecolare di malattia rara scheletrica
- o Età uguale o superiore ai 12 anni
- o Soggetti che non abbiano subito interventi chirurgici nei sei mesi precedenti l'inizio dell'arruolamento dello studio

#### ¬ Criteri di esclusione:

- Soggetti in corso di definizione diagnostica
- o Età inferiore ai 12 anni
- o Soggetti che hanno subito interventi nei sei mesi precedenti l'inizio dell'arruolamento
- o Soggetti che abbiano riportato fratture o lesioni muscolo-scheletriche nell'ultimo anno
- o Soggetti che non hanno sottoscritto il consenso informato allo studio

## 7. VARIABILI DA RILEVARE E FONTE

Le variabili analizzate saranno:

#### ¬ Informazioni generali:

- o Dati socio-demografici: età (in anni), sesso alla nascita, livello di istruzione, attività praticate nel tempo libero
- o Dati clinici: altezza, peso, limitazioni, deformità, autonomia nel cammino (quando concesso), eventuale utilizzo di ausili per la deambulazione, terapie farmacologiche, etc.
- o Dati genetici: presenza/assenza mutazione, gene, etc.
- o Dati genealogici: familiarità, ereditarietà

## ¬ Valutazione delle capacità fisiche, psicologiche, sociali e della qualità di vita:





- o Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM): questionario self-report a 34 item, versione italiana, sviluppato per misurare il cambiamento nella salute mentale secondo quattro domini (benessere soggettivo, problemi/sintomi, funzionamento e rischio) sia negli adulti sia negli adolescenti (vedi CRF)[13].
- o Pediatric Outcomes Data Collection Instrument (PODCI): questionario self-report a 83 item, versione italiana, sviluppato per misurare la funzionalità e il benessere in bambini e adolescenti con disordini dell'apparato muscolo-scheletrico, valutando sei scale (funzionalità arto superiore, mobilità, sport e attività fisica, dolore, felicità, e funzionamento globale) (vedi CRF) [14].
- o EuroQol 5-dimensions 5-levels (EQ-5D-5L): questionario generico per la valutazione della qualità della vita, versione italiana, secondo cinque dimensioni (mobilità, cura di sé, attività quotidiane, dolore/fastidio e ansia/depressione) e una scala 0-100 (vedi CRF)[15].
- o Rosenberg Self-Esteem Scale (RSES): scala composta da 10 item che richiede ai partecipanti di indicare il loro livello di accordo con una serie di affermazioni su sé stessi (vedi CRF)[16,17].

## Valutazione delle funzionalità motorie e strutture corporee tramite sensori inerziali indossabili e pedana stabilometrica (Inertial Motion Units-IMU) e parametri fisiatrici:

- o Movimenti articolari massimi, minimi ed ampiezza del movimento del torso ed arti superiori, includendo le spalle e polsi (IMU).
- o Valutazione dell'equilibrio in piedi a partire dallo spostamento del baricentro (pedana stabilometrica).
- o Punteggi di prestazione basati su standard internazionali.
- o Equilibrio, controllo del tronco in ortostasi e in posizione seduta, e controllo posturale tramite:
  - Scala di Berg: scala di valutazione dell'equilibrio e del rischio di caduta, costituita da 14 item, che indagano la capacità del paziente di mantenere una posizione, passare da una posizione a un'altra e eseguire un compito. Il punteggio massimo è di 56 punti che indica assenza di deficit di equilibrio e rischio di caduta basso/assente (vedi CRF) [18].
  - Scala di Tinetti: valuta le performance di equilibrio e deambulazione attraverso l'osservazione di abilità motorie di grande rilevanza nella vita quotidiana. Costituita da 16 items e un punteggio massimo pari a 28 (vedi CRF) [19].
  - Tampa Scale: questionario di tipo self-reporting, validato in italiano, che ha lo scopo di valutare le convinzioni sul dolore e la paura del movimento correlati al dolore in soggetti con disturbi muscoloscheletrici. Consta di 13 item e 2 sottoscale, evitamento dell'attività e focus somatico. Il punteggio può così variare da un minimo di 13 ad un massimo di 52. Dove 13 corrisponde ad assenza di chinesiofobia e 52 chinesiofobia grave (vedi CRF) [20].





#### 8. TEMPISTICA

Lo studio avrà una durata di 12 mesi coerentemente con la timeline indicata in Figura 1.



Figura 1. Timeline Pa\$

## 9. ANALISI STATISTICA

La numerosità prevista è di 8 partecipanti. Le variabili continue saranno espresse come media ± deviazione standard (SD) e mediana e range (interquartile, IQR), mentre le variabili dicotomiche o ordinali saranno espresse come percentuali e intervallo di confidenza al 95% (CI). Tenendo conto dell'esiguità della casistica, il confronto dei parametri derivanti dalle valutazioni strumentali e dei punteggi ottenuti dalla somministrazione dei questionari e delle scale sarà effettuato con test statistici non parametrici. Tali analisi verranno effettuate da biostatistici dell'Istituto Ortopedico Rizzoli.

Una definizione esatta delle future analisi dipende direttamente dalla disponibilità e dalla tipologia dei dati e dalla loro completezza.

#### 10. PROCEDURA DI ARRUOLAMENTO

Al fine di garantire la maggiore visibilità possibile allo studio e favorire l'accesso ai potenziali soggetti interessati, esso verrà promosso:

- ¬ tramite l'attività ambulatoriale della SC Malattie Rare Scheletriche,
- via piattaforme social dell'IRCCS Istituto Ortopedico Rizzoli,
- ¬ in collaborazione con UNIAMO-FIMR Federazione Italiana Malattie Rare,
- ¬ in collaborazione con le associazioni dei pazienti.

I pazienti candidabili verranno inseriti nello studio dopo aver fornito un consenso informato scritto. Nessuna raccolta dati e procedura/analisi verrà effettuata prima della firma del consenso.

## 11. RACCOLTA DATI

Per ogni paziente inserito nello studio verrà compilata la scheda raccolta dati (CRF-Scheda Raccolta Dati). I dati, pseudonimizzati, verranno collezionati su piattaforma REDcap e quindi aggregati in un unico dataset da cui verranno effettuate le analisi statistiche.

## 12. PRINCIPI ETICI

Il protocollo di ricerca e i relativi documenti saranno inviati prima di iniziare lo studio alle autorità competenti e al comitato etico per la sua approvazione.





Lo sperimentatore responsabile assicurerà che lo studio venga condotto in accordo alla Dichiarazione Helsinki nella sua versione più aggiornata (Fortaleza, Ottobre 2013), nonché con tutta la normativa nazionale ed internazionale applicabile alla ricerca clinica.

Il protocollo è stato scritto e lo studio sarà condotto secondo i principi delle ICH-GCP (rif: http://www.emea.eu.int/pdfs/human/ich/013595en.pdf).

#### 13. CONSENSO INFORMATO

Tutti i pazienti saranno informati, dallo sperimentatore, degli obiettivi dello studio, dei possibili rischi e benefici che deriveranno dalla partecipazione allo studio.

Lo sperimentatore informerà il paziente che è libero di rifiutare la partecipazione allo studio e che può ritirare il consenso in qualsiasi momento e per qualsiasi ragione.

I pazienti saranno inoltre informati sulla riservatezza dei loro dati personali; i dati dei pazienti arruolati nello studio potranno essere rivisti, ai fini dello studio, oltre che dallo sperimentatore, anche da altri individui autorizzati e comunque sempre in accordo alle norme vigenti di protezione dei dati personali e sensibili. La procedura di ottenimento del consenso informato deve essere conforme alle linee guida ICH-GCP. Ciò significa che "il modulo di consenso informato scritto deve essere firmato e datato personalmente dal

paziente o dal rappresentante legale del paziente". Lo sperimentatore sottolineerà che la partecipazione è volontaria e che al paziente è consentito ritirarsi

dallo studio in qualsiasi momento senza che questo pregiudichi le sue successive cure assistenziali.

#### 14. PRIVACY

Tutti i pazienti inclusi nello studio saranno identificati con un codice alfanumerico, in modo che i dati sensibili saranno resi pseudoanonimi e utilizzati nel rispetto della normativa in vigore in materia di privacy. I dati verranno conservati dallo sperimentatore per il tempo necessario alla produzione scientifica.

Al fine di garantire la riservatezza dei dati delle sperimentazioni cliniche come disposto dalla normativa nazionale ed europea applicabile, i dati saranno accessibili solo al promotore dello studio e i suoi designati, per le procedure di monitoraggio/auditing, allo sperimentatore e i collaboratori, e al Comitato etico del centro in cui viene condotta la ricerca e alle autorità sanitarie preposte.

Lo sperimentatore e l'Istituto consentiranno l'accesso ai dati e alla documentazione di origine per il monitoraggio, l'audit, la revisione del Comitato etico e le ispezioni dell'Autorità sanitaria, ma conservando riservatezza dei dati personali in accordo alla normativa vigente.

#### 15. REPORT FINALE E PUBBLICAZIONE DEI RISULTATI

Il responsabile dello studio, si impegna a produrre il report finale, pubblicare tutti i dati raccolti come descritto nel protocollo e a garantire che i dati siano riportati responsabilmente e coerentemente.

In particolare, la pubblicazione dei dati derivanti dal presente studio avverrà indipendentemente dai risultati ottenuti.

La trasmissione o diffusione dei dati, per il tramite di pubblicazioni scientifiche e/o di presentazione a congressi convegni e seminari, avverrà esclusivamente a seguito dell'elaborazione meramente statistica degli stessi, o comunque in forma assolutamente anonima

#### 16. FINANZIAMENTO

Lo studio è finanziato dalla donazione effettuata dalla The King Baudouin Foundation United States (KBFUS).





#### 17. BIBLIOGRAFIA

- 1. Committee for Medicinal Products for Human Use. (2013). European Medicines Agency. European Public Assessment Report: procedure no. EMEA/H/C/000471/II/0082: Aripiprazole. 2013. 12-2-2013.
- 2. Institute of Medicine (US) Committee on Accelerating Rare Diseases Research and Orphan ProductDevelopment. Rare Diseases and Orphan Products: Accelerating Research and Development; Field, M. J., Boat, T. F., Eds.; The National Academies Collection: Reports funded by National Institutes of Health; National Academies Press (US): Washington (DC), 2010.
- 3. UNIAMO (**2022**). MonitoRare. Ottavo Rapporto sulla condizione della persona con Malattia Rara in Italia. Anno 2022
- 4. Cornaglia Ferraris, P. [Adventure therapy: principles, practice, perspectives.]. Recenti Prog Med 2018, 109 (10), 487–493. https://doi.org/10.1701/3010.30086.
- 5. MacLachlan M. Sailing as an Intervention. In: MacLachlan M, editor. Maritime Psychology: Research in Organizational & Health Behavior at Sea. Cham: Springer International Publishing; **2017**. <a href="https://doi.org/10.1007/978-3-319-45430-6\_10">https://doi.org/10.1007/978-3-319-45430-6\_10</a>
- 6. Thompson T, Lamont-Robinson C, Williams V. At sea with disability! Transformative learning in medical undergraduates voyaging with disabled sailors. Med Educ. **2016** Aug;50(8):866–79. https://doi.org/10.1111/medu.13087
- 7. Recio AC, Becker D, Morgan M, Saunders NR, Schramm LP, McDonald JWI. Use of a Virtual Reality Physical Ride-On Sailing Simulator as a Rehabilitation Tool for Recreational Sports and Community Reintegration: A Pilot Study. American Journal of Physical Medicine & Rehabilitation. 2013 Dec;92(12):1104. https://doi.org/10.1097/PHM.00000000000000012
- 8. Tracey, D.; Gray, T.; Truong, S.; Ward, K. Combining Acceptance and Commitment Therapy With Adventure Therapy to Promote Psychological Wellbeing for Children At-Risk. *Front Psychol* **2018**, 9, 1565. <a href="https://doi.org/10.3389/fpsyg.2018.01565">https://doi.org/10.3389/fpsyg.2018.01565</a>.
- 9. Capurso, M.; Borsci, S. Effects of a Tall Ship Sail Training Experience on Adolescents' Self-Concept. International Journal of Educational Research 2013, 58, 15–24. https://doi.org/10.1016/j.ijer.2013.01.004.
- 10.Gill, E.; Goldenberg, M.; Starnes, H.; Phelan, S. Outdoor Adventure Therapy to Increase Physical Activity in Young Adult Cancer Survivors. *J Psychosoc Oncol* **2016**, 34 (3), 184–199. https://doi.org/10.1080/07347332.2016.1157718.
- 11.Zebrack, B.; Kwak, M.; Sundstrom, L. First Descents, an Adventure Program for Young Adults with Cancer: Who Benefits? Support Care Cancer 2017, 25 (12), 3665–3673. <a href="https://doi.org/10.1007/s00520-017-3792-7">https://doi.org/10.1007/s00520-017-3792-7</a>.
- 12. Aprile I, Iacovelli C, Iuvone L, Imbimbo I, Cruciani A, Pecchioli C, et al. Use of a Virtual-Technological Sailing Program to Prepare Children With Disabilities for a Real Sailing Course: Effects on Balance and Quality of Life. J Child Neurol. 2016 Jul;31(8):1074–80. https://doi.org/10.1177/0883073816638756
- 13. Palmieri, G.; Reitano, F. La valutazione degli esiti degli interventi psicologici e il questionario CORE-OM. *RIVISTA SPERIMENTALE DI FRENIATRIA* **2014**, No. 2014/1. https://doi.org/10.3280/RSF2014-001008.
- 14.Trisolino, G.; Stallone, S.; Zarantonello, P.; Evangelista, A.; Boarini, M.; Faranda Cordella, J.; Lerma, L.; Veronesi, L.; Guerra, C. C.; Sangiorgi, L.; Di Gennaro, G. L.; Toniolo, R. M. Translation and Cross-Cultural Adaptation of the Pediatric Outcomes Data Collection Instrument into the Italian Language. *Children* **2022**, 9 (6), 853. <a href="https://doi.org/10.3390/children9060853">https://doi.org/10.3390/children9060853</a>.
- 15. Finch, A. P.; Meregaglia, M.; Ciani, O.; Roudijk, B.; Jommi, C. An EQ-5D-5L Value Set for Italy Using Videoconferencing Interviews and Feasibility of a New Mode of Administration. *Social Science & Medicine* 2022, 292, 114519. https://doi.org/10.1016/j.socscimed.2021.114519.
- 16.Rosenberg M. Society and the Adolescent Self-Image. Princeton: Princeton University Press





## 1965. https://doi.org/10.1515/9781400876136

- 17. Prezza, M.; Trombaccia, F. R.; Armento, L. La Scala Dell'autostima Di Rosenberg: Traduzione e Validazione Italiana. [The Rosenberg Self-Esteem Scale: Italian Translation and Validation.]. *Giunti Organizzazioni Speciali* 1997, 223, 35–44.
- 18.Ottonello M, Ferriero G, Benevolo E, Sessarego P, Dughi D. Psychometric evaluation of the italian version of the berg balance scale in rehabilitation inpatients. *Europa Medicophysica*. **2003**;39(4):181-189.<a href="https://www.proquest.com/scholarly-journals/psychometric-evaluation-italian-version-berg/docview/204123075/se-2">https://www.proquest.com/scholarly-journals/psychometric-evaluation-italian-version-berg/docview/204123075/se-2</a>.
- 19.Tinetti ME. Performance-oriented assessment of mobility problems in elderly patients. *J Am Geriatr Soc.* **1986**;34(2):119-126. <a href="https://doi.org/10.1111/j.1532-5415.1986.tb05480.x">https://doi.org/10.1111/j.1532-5415.1986.tb05480.x</a>
- 20. Monticone M, Giorgi I, Baiardi P, Barbieri M, Rocca B, Bonezzi C. Development of the Italian version of the Tampa Scale of Kinesiophobia (TSK-I): cross-cultural adaptation, factor analysis, reliability, and validity. Spine (Phila Pa 1976). 2010;35(12):1241-1246. https://doi.org/10.1097/BRS.0b013e3181bfcbf6
- 21. Federici, S.; Meloni, F.; Mancini, A.; Lauriola, M.; Olivetti Belardinelli, M. World Health Organisation Disability Assessment Schedule II: Contribution to the Italian Validation. *Disability and Rehabilitation* **2009**, 31 (7), 553–564. https://doi.org/10.1080/09638280802240498.
- 22. Maini, M.; Nocentini, U.; Prevedini, A.; Giardini, A.; Muscolo, E. An Italian Experience in the ICF Implementation in Rehabilitation: Preliminary Theoretical and Practical Considerations. *Disability and Rehabilitation* 2008, 30 (15), 1146–1152. https://doi.org/10.1080/09638280701478397.
- 23.Hernandez-Lazaro, H.; Mingo-Gómez, M. T.; Ceballos-Laita, L.; Medrano-de-la-Fuente, R.; Jimenez-del Barrio, S. Validation of the International Classification of Functioning, Disability, and Health (ICF) Core Sets for Musculoskeletal Conditions in a Primary Health Care Setting from Physiotherapists' Perspective Using the Delphi Method. *Disability and Rehabilitation* **2023**, *45* (15), 2458–2468. https://doi.org/10.1080/09638288.2022.2096128.

# Ready to Sail: Feasibility Study on the Impact of Sailing as Ergotherapy in Patients with Rare Skeletal Diseases

## Acronym:

PaS

#### **Sponsor and Address:**

IRCCS - Rizzoli Orthopedic Institute Via di Barbiano 1/10, 40136 Bologna, Italy

#### **Protocol Version and Date:**

Version 1.1, dated March 22, 2024

## **Coordinating Center:**

Rare Skeletal Diseases Department – IRCCS Rizzoli Orthopedic Institute

## **Principal Investigator:**

Dr. Luca Sangiorgi

Phone: +39 051 6366342 Email: luca.sangiorgi@ior.it

## Other Participating Institutions:

- Physical Medicine and Rehabilitation Unit 1 IRCCS Rizzoli Orthopedic Institute
- Physical Medicine and Rehabilitation Unit 2 IRCCS Rizzoli Orthopedic Institute
- Motion Analysis Laboratory IRCCS Rizzoli Orthopedic Institute
- MARINANDO ODV/MARINANDO 2.0 APS ASD, Rimini

Methodology: Single-center interventional pilot study

Type: Non-profit

## **Funding Source:**

The King Baudouin Foundation United States (KBFUS), Project Code: 2024/731019

## **Principal Investigator's Declaration:**

I confirm that I have read the protocol and agree to conduct this study in accordance with ICH-GCP guidelines, the protocol specifications, and applicable regulations.

Dr. Luca Sangiorgi (Signature)

#### **Table of Contents**

- 1. Rationale
- 2. Study Objectives
- 3. Study Design
- 4. Expected Results
- 5. Study Setting

- 6. Study Population
- 7. Variables to Be Collected and Sources
- 8. Study Timeline
- 9. Statistical Analysis
- 10. Recruitment Procedure
- 11. Data Collection
- 12. Ethical Principles
- 13. Informed Consent
- 14. Privacy
- 15. Final Report and Publication of Results

#### 1. Rationale

Rare diseases are defined as conditions that affect a small number of individuals and are characterized by chronic debilitating symptoms 【1】. According to WHO estimates, approximately 300 million people globally, 27–36 million in Europe, and 2.1–3.5 million in Italy are affected by rare diseases 【2,3】. These conditions significantly impact individuals, families, and the broader social and healthcare systems.

To address the challenges arising from the rarity of such conditions, several measures have been implemented at both the community and national levels [3]. In Italy, the 2013–2016 National Plan for Rare Diseases and the more recent "Rare Diseases Consolidated Act" (Law No. 175/2021) emphasize the development of integrated strategies centered on the needs of patients and their families. These strategies aim to improve diagnostic and therapeutic pathways, promote timely diagnoses, ensure access to innovative therapies, and empower patients and their families.

Adventure Therapy (AT) is an experiential treatment approach that has demonstrated effectiveness in enhancing self-esteem, autonomy, and social skills in individuals with rare, chronic, or disabling conditions [4]. By facilitating interaction among individuals, groups, and nature, it promotes holistic physical, cognitive, emotional, and social rehabilitation. Sailing, as a form of Adventure Therapy, is particularly valued for fostering enjoyment, inclusion, and participation [5-7]. Studies highlight the benefits of such emotionally engaging and recreational experiences, especially for patients with chronic, genetic, metabolic, or oncological diseases [8-11].

From a rehabilitative perspective, sailing activities positively impact physical functioning and participation, as defined by the International Classification of Functioning (WHO, 2001). Participants report improved physical capabilities and enhanced life satisfaction [7,12].

This study aims to assess the feasibility of using sailing as ergotherapy to improve physical, cognitive, and social abilities in patients with rare skeletal diseases.

## 2. Study Objectives

## **Primary Objective:**

To evaluate the feasibility of implementing a nautical ergotherapy program for improving physical, psychological, and social capabilities in individuals with rare skeletal diseases.

## **Secondary Objectives:**

- Assess changes in perceived safety and ability to perform movements.
- Measure improvements in self-worth and capabilities.
- Evaluate changes in quality of life.
- Identify a standardized set of functional parameters and rehabilitation exercises.

## 3. Study Design

**Type**: Single-center, interventional pilot study.

#### Phases:

- 1. Recruitment (Phase 1): Promotion, participant enrollment, and baseline evaluation (T0).
- 2. **Pre-boarding (Phase 2)**: Training sessions on nautical activities.
- 3. Sailing (Phase 3): Intervention with pre-activity (T1) and post-activity evaluations (T2).
- 4. Follow-up (Phase 4): Final evaluation three months post-intervention (T3).

## **Assessment Tools:**

- Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM)
- Pediatric Outcomes Data Collection Instrument (PODCI)
- EuroQol 5-Dimensions (EQ-5D)
- Rosenberg Self-Esteem Scale (RSES)
- Tinetti Scale
- Berg Balance Scale
- Tampa Scale

Each phase and its corresponding activities and assessments are detailed in Table 1.

Table 1: Study Phases and Activities

| Phase | Activities | Assessment Tools |
|---|---|---|
| Phase 1 | Recruitment, informed consent, and baseline | CORE-OM, PODCI, EQ-5D, RSES, |
| riiase 1 | evaluation (T0) | Tinetti Scale, Berg Scale |
| Phase 2 | Training sessions on sailing principles and practices | Not applicable |
| | Pre-activity evaluation (T1), sailing intervention, | CORE-OM, PODCI, EQ-5D, RSES, |
| Phase 3 | debriefing, and post-activity evaluation (T2) | Tinetti Scale, Berg Scale, Inertial |
| | | Movement Units (IMU) |

| | | | CORE-OM, PODCI, EQ-5D, RSES, |
|---|---|---|---|
| F | Phase 4 | Follow-up evaluation (T3) | Tinetti Scale, Berg Scale, Inertial |
| | | | Movement Units (IMU) |

I will continue translating the remaining sections (Expected Results, Study Setting, Study Population, etc.) in the next response.

## 4. Expected Results

The expected outcomes of the sailing intervention are categorized as follows:

## **Short-Term Outcomes (Pre- and Post-Intervention Evaluation)**:

## Physical Benefits:

- o Increased muscle strength and endurance.
- o Improved muscle tone and proprioception (body awareness).
- o Enhanced posture control and coordination.
- Strengthening of stabilizing muscles.

## Psychological Benefits:

- o Greater self-awareness and confidence.
- Acquisition of new skills.
- Reinforcement of trust in one's abilities.
- o Improved socialization skills.

#### Medium-Term Outcomes (3-Month Follow-Up):

## Physical Benefits:

- o Consolidation of muscle strength, endurance, and tone.
- o Stabilization of improved posture control and coordination.

## Psychological Benefits:

- Enhanced ability to face challenges.
- Sustained self-awareness and confidence.
- o Stabilization of social skills and participation.

## 5. Study Setting

The study activities will be conducted across the following locations:

## • Recruitment, Informed Consent, and Follow-Up:

Rare Skeletal Diseases Unit, IRCCS Rizzoli Orthopedic Institute, Bologna.

## • Training:

Conducted online via GoToMeeting platform.

## Sailing Activities and Accommodation:

- Marina di Ravenna Tourist Harbor (Marinara), in collaboration with MARINANDO ODV.
- o Palazzo Manzoni, San Zaccaria, for accommodation and additional activities.

#### 6. Study Population

#### Sample Size:

The study is a feasibility pilot, targeting a maximum of 8 participants due to the rarity of the condition.

#### **Inclusion Criteria:**

- Individuals of any gender aged 12 years or older.
- Clinical or molecular diagnosis of a rare skeletal disease.
- No surgical procedures within six months prior to recruitment.

#### **Exclusion Criteria:**

- Undetermined diagnosis.
- Age below 12 years.
- Fractures or musculoskeletal injuries within the past year.
- Declined to provide written informed consent.

#### 7. Variables to Be Collected and Sources

#### **General Information:**

- **Sociodemographic Data**: Age, sex, education level, recreational activities.
- **Clinical Data**: Height, weight, physical limitations, deformities, use of assistive devices, and current pharmacological treatments.
- **Genetic Data**: Mutation presence affected gene(s).
- **Genealogical Data**: Family history and inheritance patterns.

## **Functional, Psychological, and Social Evaluations:**

- **CORE-OM**: Measures mental health across subjective well-being, symptoms, functioning, and risk domains.
- **PODCI**: Evaluates functionality and well-being in pediatric musculoskeletal disorders using six scales.
- **EQ-5D-5L**: Assesses quality of life across mobility, self-care, daily activities, pain/discomfort, and anxiety/depression.
- RSES: Assesses self-esteem through 10 items.
- Motor and Balance Assessment: Using wearable Inertial Motion Units (IMUs), stabilometric platforms, and physiotherapy scales such as the Tinetti and Berg scales.

#### 8. Study Timeline

The study will span 12 months. Specific phases and activities are outlined in the timeline provided in Figure 1 of the protocol.



Figure 1. Pa\$ Timeline

## 9. Statistical Analysis

Continuous variables will be expressed as mean ± standard deviation and median (interquartile range). Dichotomous or ordinal variables will be presented as percentages with 95% confidence intervals. Due to the small sample size, non-parametric tests will be used for statistical comparisons. Analyses will be conducted by biostatisticians at IRCCS Rizzoli Orthopedic Institute.

#### 10. Recruitment Procedure

To ensure maximum visibility and accessibility, the study will be promoted via:

- Outpatient services of the Rare Skeletal Diseases Department.
- IRCCS Rizzoli Orthopedic Institute's social media platforms.
- UNIAMO-FIMR Italian Federation for Rare Diseases.
- Collaboration with patient associations.

Eligible participants will be enrolled after providing written informed consent. No data collection or analysis will occur before obtaining consent.

#### 11. Data Collection

For each participant, a Case Report Form (CRF) will be compiled. Data will be pseudonymized, stored on the REDCap platform, and aggregated into a single dataset for statistical analysis.

#### 12. Ethical Principles

The protocol and related documents will be submitted to competent authorities and an ethics committee for approval prior to study initiation. The study will comply with the latest version of the Declaration of Helsinki (Fortaleza, 2013) and applicable national and international regulations.

## 13. Informed Consent

Participants will receive detailed information about the study's objectives, risks, and benefits. Written informed consent must be obtained, with participants free to withdraw at any time without impacting on their future care.

## 14. Privacy

Participants' personal data will be pseudonymized and handled per current national and European privacy regulations. Access to data will be restricted to authorized personnel, including the sponsor, investigators, and ethics committees.

## 15. Final Report and Publication of Results

The study's results will be published regardless of the outcomes, ensuring anonymity and compliance with ethical standards. Findings will be disseminated through scientific journals, conferences, and seminars.